CLINICAL TRIAL: NCT00399243
Title: 4mg StatDose Imitrex for Acute Treatment of Cluster Headache
Brief Title: Sumatriptan 4 mg Statdose in the Acute Treatment of Cluster Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diamond Headache Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Frederick Freitag, D.O., Diamond Headache Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHC08
Record Dates: First submitted 2006-11-12; First posted 2006-11-14 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Episodic Cluster Headache; Chronic Cluster Headache
Keywords: cluster headache; sumatriptan
MeSH Terms: conditions — Cluster Headache | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sumatriptan 4mg Statdose injection — 4mg Sumatriptan Statdose injection for use as acute therapy in a cluster headache. Consistency of response in three attacks will be measured

SUMMARY:
This study's hypothesis is the 4mg StatDose sumatriptan is effective for the acute treatment of cluster headache and provides good safety and tolerability across multiple doses of the study medication as well as across multiple attacks of cluster headache. This study seeks to determine the safety and efficacy of the commercially available 4mg StatDose formulation of sumatriptan as an acute treatment of cluster headache. Patients are allowed to use repeated dose of the study medication for a given headache if they have had a partial response to the first dose. They may treat up to 3 attacks of cluster headache with the study medication. Safety assessment will be through adverse event reporting and physical examination. Patients with both episodic cluster headache as well as chronic cluster headache will be studied. Patients must either not have started preventive treatment for cluster headache or be on a stable dose of preventive medication.

DETAILED DESCRIPTION:
This is an open label trial of sumatriptan 4 mg using the StatDose injector system for the treatment of acute attacks of cluster headache.

Patient entering the trial must either be in the first 3 weeks of an episodic cluster headache cycle or have chronic cluster headache. Patients with episodic cluster headache may have not begun taking preventive medications at the time of study or must be on a stable regimen of preventive medications. Patients with chronic cluster headache must be on a stable regimen of preventive medications.

Patients must be in good health with no contraindications to the use of sumatriptan such as either having or having increased risk factors for CAD or CVD. They may not take during the time of the study preventive medications that are 5HT1B/1D agonists. Episodic use of triptans, ergotamine, or dihydroergotamine is permitted provided they are not used within 24 hours of use of the study medication.

Patients will be required to treat 3 acute attacks of cluster headache with the study medication or to use more than 1 dose of study medication to fully treat an individual attack of cluster headache with a maximum of 3 doses of the study medication within a 24 hour time frame.

Efficacy of the study medication will be determined from diary data collected. Safety data will be determined by adverse events reported by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 years and 65 years of age.
* Subject is male or female. If female the subject is:
* non-childbearing potential or,
* child-bearing potential, has a negative pregnancy test at screen, and agrees to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug (a minimum of 10 hours); or,
* Female sterilization; or,
* Sterilization of male partner; or,
* Implants of levonorgestrel; or,
* Injectable progestogen; or,
* Oral contraceptive (combined or progestin only) or,
* Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year; or,
* Double barrier method; (2 physical barriers or 1 physical barrier plus spermicide).
* Subject has a diagnosis of cluster headache (IHS).
* Subject has at least 1 previous cycle of cluster headache if episodic or has been in chronic cluster headache for at least 6 months.
* Subject taking any medication for chronic cluster headache prevention has been on a stable regimen for at least 1 month prior to screening.
* Subjects with episodic cluster headache have a history of continuing to have cluster headaches at least once every other day during the first three weeks of treatment with preventive medications.
* Subject is able and willing to give written informed consent to participate in the study.
* Subject who have used 6 mg StatDose Imitrex for the treatment of cluster headache must have a history of responding to treatment with this in at least 1 out every 3 attacks.

Exclusion Criteria:

* Subject has confirmed or suspected ischemic heart disease, Prinzmetal's angina, or signs/symptoms consistent with any of the above.
* Subject has cardiac arrhythmias requiring medication or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion contraindicates participation in this study.
* Subject has a history of congenital heart disease.
* Subject has a history of cerebrovascular pathology including stroke.
* The subject, in the investigator's opinion, is likely to have unrecognized cardiovascular disease.
* Subject has evidence or history of ischemic abdominal syndromes or peripheral vascular disease.
* Subject has uncontrolled hypertension at screening.
* Subject has a history of epilepsy or structural brain lesions which lowers the convulsive threshold.
* Subject has a history of impaired hepatic or renal function.
* Subject is currently taking a monoamine oxidase inhibitor (MAO) or has taken a MAOI within the 2 weeks prior to screen
* Subject is currently taking an ergotamine-containing or ergot-type cluster headache preventive medication like ergotamine tartrate or methylergonovine.
* Subject has hypersensitivity or contraindication to the use of sumatriptan, any of its components, or any other 5-HT1B1D receptor agonist.
* Subject is pregnant, actively trying to become pregnant or breast-feeding
* Subject is of childbearing potential and not using adequate contraceptive measures.
* Subject has evidence of alcohol or substance abuse within the last year which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results.
* Subject has any concurrent medical or psychiatric condition that, in the investigator's opinion, may affect the interpretation of efficacy and safety date or which otherwise contraindicates participation in a clinical trial.
* Subject has participated in an investigational drug trial within the previous four weeks.
* Subject is unable or unwilling to self administer subcutaneously administered Imitrex.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy parameters will be the percentage of cluster headache attacks that result in the cluster headache pain being reduced to mild or none following a single dose of 4 mg subcutaneous sumatriptan at 15 minutes and at 30 minutes. | 15 minutes and 30 minutes

SECONDARY OUTCOMES:
The time meaningful relief of cluster headache. | Meaningful Relief
The percentage of attacks that produce a pain free response to a single dose of sumatriptan 4 mg subcutaneous at 15 minutes, 30 minutes and at 1 hour. | 30 minutes and 1 Hour
The percentage of attacks of migraine that result in resolution of all associated symptoms of cluster headache present at the time of treatment with the study medication as well as achieving a pain free response within 1hour. | 1 hour
The number of patients reporting adverse effects to study medication, the type of adverse event reported and the percentage of attacks that are associate with the adverse effect. | Length of study
The percentage of patients who achieve pain reduced to mild or none at 15 minutes or at 30 minutes respectively for all three treated headache attacks. | 15 minutes and 30 minutes
The percentage of patients who achieve pain reduced to mild or none at 15 minutes or at 30 minutes respectively for two out of three treated headaches. | 15 minutes and 30 minutes
The percentage of patients who become pain free at 15 minutes or 30 minutes or at 1 hour respectively or at any combination of the three time points for all three headache attacks. | 15 minutes, 30 minutes, and 1 hour
Patient evaluation of subcutaneous sumatriptan 4 mg regarding satisfaction with their treatment using the PPMQR assessment. | End of treatment
The percentage of attacks in which the pain was reduced to moderate or mild and for which the patient took a second and or a third dose of the study medication. | Length of study
The percentage of attacks in which the patient became pain free at or before 1 hour and experienced a recurrence of cluster headache and in which a second or third dose of study medication was taken. | 1 hour
The percentage of cluster headaches in which the patient became free at or before 1 hour and experienced a recurrence of cluster headache. | 1 hour
The mean time to meaningful pain relief across three treated headache attacks. | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Seymour Diamond, MD, Principal Investigator — Diamond Headache Clinic
Locations (1):
- Diamond Headache Clinic, Chicago, Illinois, United States